CLINICAL TRIAL: NCT01646593
Title: An Open-label Expanded Access Program of Regorafenib in Patients With Gastrointestinal Stromal Tumors (GIST) After Disease Progression on or Intolerance to Imatinib and Sunitinib
Brief Title: Regorafenib in Subjects With Gastrointestinal Stromal Tumors (GIST) Who Have Progressed After Standard Therapy
Status: No longer available | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Other Study IDs: 16339
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506) — 160 mg BAY73-4506, 3 weeks on drug, 1 week off

SUMMARY:
The objective of the trial is to provide regorafenib to subjects diagnosed with metastatic and / or unresectable GIST who have progressed after standard therapy.

Selected additional safety information on regorafenib will be collected and progression-free survival (PFS) will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >= 18 years of age
* Subjects with histologically confirmed metastatic and / or unresectable GIST
* At least imatinib and sunitinib as prior treatment regimens with progression on or intolerance to imatinib and sunitinib
* Adequate bone marrow, liver and renal function
* Women of childbearing potential and men must agree to use adequate contraception before entering the program until at least 8 weeks after the last study drug administration. The investigator or a designated associate is requested to advise the subject on how to achieve adequate birth control. Adequate contraception is defined in the study as any medically recommend method (or combination of methods) as per standard of care.

Exclusion Criteria:

* Prior treatment with regorafenib
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting study drug
* Pregnant or breast-feeding subjects. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of study drug.
* Congestive heart failure >= New York Heart Association (NYHA) class 2
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
* Myocardial infarction less than 6 months before start of study drug
* Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension (Systolic blood pressure > 140 mmHg or diastolic pressure > 90 mmHg despite optimal medical management)
* Pleural effusion or ascites that causes respiratory compromise (National Cancer Institute Common terminology criteria for adverse events [NCI-CTCAE] v. 4.0 Grade >= 2 dyspnea)
* Ongoing infection NCI-CTCAE v. 4.0 Grade > 2
* Known history of human immunodeficiency virus (HIV) infection
* Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy
* Subjects with seizure disorder requiring medication
* History of organ allograft
* Subjects with evidence or history of any bleeding diathesis, irrespective of severity
* Any hemorrhage or bleeding event NCI-CTCAE v. 4.0 Grade >= 3 within 4 weeks prior to the start of study medication
* Non-healing wound, ulcer, or bone fracture
* Renal failure requiring hemo- or peritoneal dialysis
* Dehydration NCI-CTCAE v. 4.0 Grade >= 1
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Known hypersensitivity to the study drug, study drug class, or excipients in the formulation
* Any illness or medical conditions that are unstable or could jeopardize the safety of the subject and his / her compliance in the study
* Interstitial lung disease with ongoing signs and symptoms
* Persistent proteinuria of NCI-CTCAE v. 4.0 Grade 3 (> 3.5 g/24 hours)
* Subjects unable to swallow oral medications
* Any malabsorption condition
* Unresolved toxicity higher than NCI-CTCAE v. 4.0 Grade 1 (excluding alopecia, anaemia,and hypothyroidism) attributed to any prior therapy / procedure
* Concomitant participation or participation in another therapeutic trial with investigational new drugs within 30 days or 5 drug half-lives (if drug half life in subjects is known), whichever is shorter
* If any other approved tyrosine kinase inhibitor was given within 1 week or a minimum of 5 drug half-lives whichever is longer (i.e. within 7 days for imatinib, or within 10 days for sunitinib)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer